CLINICAL TRIAL: NCT05123313
Title: Medication Use and Quality of Life Among Older People
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Carina Lundby, Postdoctoral Researcher, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ODIN-1
Record Dates: First submitted 2021-10-27; First posted 2021-11-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Quality of Life; Reduction, Harm
Keywords: Deprescribing; Polypharmacy; Shared decision-making; Guideline
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will not receive a series of consultations with their general practitioner. Controls will receive baseline measurements and follow-up measurements 3 months and 6 months following baseline measurements.
- Intervention group (Experimental): The intervention will comprise a series of consultations between the patient and general practitioner (at least three), where the patient and general practitioner will continuously adjust the patient's medication according to the patient's goals, needs, and preferences. Interventions will receive baseline measurements and follow-up measurements 3 months and 6 months following baseline measurements.
  Interventions: Behavioral: Deprescribing intervention

INTERVENTIONS:
Behavioral: Deprescribing intervention — The intervention is comprised of a minimum of three consultations with a general practitioner (GP), where adjustment of the patient's medication is made according to the patient's preference, goals and needs
  Consultation 1: Patient and GP discuss how the patient feels about their medical treatment, and the GP provides the patient with written material for the patient to prepare prior to the next consultation.
  Consultation 2: A clinical pharmacist have beforehand examined the patient's medication list and provided suggestions to the GP on which drugs can be deprescribed. The patient and GP discuss the patient's preferences and initiate deprescribing initiatives aligned with the patient's priorities.
  Consultation 3: Patient and GP follow up on the changes initiated and initiate new deprescribing initiatives if such can be identified. If needed, subsequent consultations (Consultation X) are planned until the patient and GP consider the patient's medical treatment optimal.
  Arms: Intervention group

SUMMARY:
This project will provide new evidence on how to optimize medication use among older people with limited life expectancy. This will be done by testing whether a patient-centered deprescribing intervention, focused on aligning medical treatment with patients' preferences, can improve quality of life among older people with limited life expectancy.

DETAILED DESCRIPTION:
In a pragmatic randomized controlled trial, this project will test whether a comprehensive and patient-centered deprescribing intervention can improve quality of life among older people with limited life expectancy. The intervention will comprise a series of consultations between the patient and general practitioner (GP) (at least three) to continuously adjust the patient's medication according to the patient's goals, needs, and preferences, thereby ensuring alignment with the patient's priorities. Thus, the purpose of this intervention is to initiate and facilitate a continued deprescribing process.

The process can be summarized in eight steps: During an initial consultation (1: Consultation 0), the GP assesses patient eligibility. If the patient would like to participate, a project nurse subsequently visits the patient at home (2: Home visit) for retrieval of informed consent as well as baseline measurements. After retrieval of informed consent, patients are randomized. Patients randomized to the control group continue with usual care (consultations with their GP when needed). Patients in the intervention group receive the intervention, comprising a series of consultations between the patient and GP (at least three). During the first intervention consultation (3: Consultation 1), the patient and GP discuss how the patient feels about their medical treatment, and the GP provides the patient with written material for the patient to prepare prior to the next consultation. The patients prepare (4: Preparation) by considering and verbalizing their goals of care and treatment preferences. Simultaneously, a clinical pharmacist examines the patient's medication list and provides suggestions to the GP on which drugs can be continued and deprescribed, respectively. During the next intervention consultation (5: Consultation 2), the patient and GP discuss the patient's preferences and initiate deprescribing initiatives aligned with the patient's priorities. During a new intervention consultation (6: Consultation 3), the patient and GP follow up on the changes initiated and initiate new deprescribing initiatives if such can be identified. If needed, subsequent intervention consultations (7: Consultation X) are planned until the patient and GP consider the patient's medical treatment optimal. A project nurse visits all patients (both patients randomized to the control and intervention group, respectively) at home 3 and 6 months after first home visit to retrieve follow-up measurements (8: Follow-ups). A project nurse retrieves medication lists at 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 80 years
* Take ≥ 8 different medications
* Have a life expectancy of <2 years, estimated via the Surprise Question ("Would you be surprised if this patient died within 1-2 years?") by the general practitioner
* have a Mini-Mental State Exam (MMSE) score of ≥18
* Are able to provide informed consent

Exclusion Criteria:

* Not able to communicate
* Does not speak and understand Danish

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HEALTH-RELATED QUALITY OF LIFE | Baseline
  Health-related quality of life will be measured using the Danish version of the Short Form 12 Health Survey Version 2 (SF-12v2).
CHANGE FROM BASLINE HEALTH-RELATED QUALITY OF LIFE AT 3 MONTHS | 3 months
  Health-related quality of life will be measured using the Danish version of the Short Form 12 Health Survey Version 2 (SF-12v2).
CHANGE FROM BASLINE HEALTH-RELATED QUALITY OF LIFE AT 6 MONTHS | 6 months
  Health-related quality of life will be measured using the Danish version of the Short Form 12 Health Survey Version 2 (SF-12v2).
HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) | Baseline
  Health-related quality of life will be measured using the Danish version of the Depression List (DL).
CHANGE FROM BASLINE HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) AT 3 MONTHS | 3 months
  Health-related quality of life will be measured using the Danish version of the Depression List (DL).
CHANGE FROM BASLINE HEALTH-RELATED QUALITY OF LIFE (DEPRESSION) AT 6 MONTHS | 6 months
  Health-related quality of life will be measured using the Danish version of the Depression List (DL).
MORTALITY | 3 months
  Mortality will be assessed through the nationwide Danish Central Person Registry (CPR).
MORTALITY | 6 months
  Mortality will be assessed through the nationwide Danish Central Person Registry (CPR).
MORTALITY | 12 months
  Mortality will be assessed through the nationwide Danish Central Person Registry (CPR).

SECONDARY OUTCOMES:
COGNITIVE FUNCTION | Baseline, 3 months and 6 months
  Cognitive function will be measured using the Danish version of the Mini-Mental State Examination Version 2 Standard Form (MMSE-2).
FUNCTIONAL LEVEL | Baseline, 3 months and 6 months
  Functional level will be measured using the Danish version of the Vulnerable Elders Survey 13 (VES-13).
HAND-GRIP STRENGTH | Baseline, 3 months and 6 months
  Hand-grip strength will be measured using a hand-grip dynamometer.
NUMBER OF MEDICATION DISCONTINUED | 3 months, 6 months and 12 months
  Number of medications discontinued will be assessed through the medication lists.
NUMBER OF MEDICATION CHANGES | 3 months, 6 months and 12 months
  Number of medication changes will be assessed through the medication lists.
HOSPITAL ADMISSIONS | 3 months, 6 months and 12 months
  Hospital admissions will be assessed through the nationwide Danish National Patient Registry.
HEALTH CARE COSTS | 3 months, 6 months and 12 months
  Health care costs will be assessed through nationwide Danish Health Care registries.
SUCCESS RATE OF THE INTERVENTION | 3 months, 6 months and 12 months
  Success rate will be assessed through persisting discontinuations and changes of medications via the medication lists.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Pottegård, Professor, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No